CLINICAL TRIAL: NCT01550562
Title: Precision™ High-Rate Sub-perception Spinal Cord Stimulation for the Treatment of Chronic Intractable Pain
Brief Title: Effects of Programming Parameters on Back Pain Relief in Subthreshold Spinal Cord Stimulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In >9 months only 1 patient enrolled. Study stopped because design was too cumbersome and subjects not willing to participate
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A7002
Record Dates: First submitted 2012-02-15; First posted 2012-03-12 (Estimated); Results first posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sham Stimulation (Placebo Comparator): Sham subthreshold spinal cord stimulation therapy
  Interventions: Device: Boston Scientific Precision Plus spinal cord stimulation therapy
- Treatment 1 (Active Comparator): subthreshold spinal cord stimulation therapy
  Interventions: Device: Boston Scientific Precision Plus spinal cord stimulation therapy
- Treatment 2 (Experimental): subthreshold spinal cord stimulation therapy
  Interventions: Device: Boston Scientific Precision Plus spinal cord stimulation therapy

INTERVENTIONS:
Device: Boston Scientific Precision Plus spinal cord stimulation therapy — Epidural spinal cord stimulation (SCS) using the Boston Scientific Precision Plus SCS system

SUMMARY:
The purpose of this study is to investigate the effects of varying programming parameters in subthreshold spinal cord stimulation therapy for pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Chronic intractable pain of the trunk and/or limbs
* Documented history of trunk and/or limb pain of at least 180 days
* Average back pain intensity of 5 or greater on a 0-10 numerical rating scale during the 7-day period prior to the Screening Visit
* Pass study site's routine psychological/psychiatric evaluation within 180 days of the Trial Lead Insertion Visit
* If taking any medications for chronic pain, must be on a stable prescription during the 14-day period prior to the Trial Lead Insertion Visit and agree to continue on the same prescription throughout study participation
* Subject is willing and able to comply with all protocol-required procedures and assessments/evaluations
* Subject is able to independently read and complete all questionnaires and/or assessments provided in English
* 18 years of age or older when written informed consent is obtained
* Subject signs a valid, Ethics Committee-approved informed consent form (ICF) provided in English

Exclusion Criteria:

* Unable to operate the PrecisionPlus™ system
* Primary source of pain is cancer-related, pelvic, visceral, angina, or migraine
* Is a high surgical risk
* Is diabetic
* Is immunocompromised
* Currently on any anticoagulant medications that cannot be discontinued during perioperative period
* Untreated major depression or untreated generalized anxiety disorder
* Diagnosed with somatoform disorder, severe personality disorder, borderline personality disorder
* Diagnosed with any major psychiatric disorder not specifically listed in previous two exclusion criterion
* Currently diagnosed with cognitive impairment that would limit subject's ability to discern differences in pain severity, complete a pain diary, perform wound care
* Current abuse of alcohol or illicit drugs
* Subject requires Magnetic Resonance Imaging (MRI) while implanted with lead(s).
* Subject is participating (or intends to participate) in another investigational drug or device clinical trial that may influence the data that will be collected for this study
* Subject has previously undergone a spinal cord stimulation trial or is already implanted with an active implantable device(s) to treat their pain (IPGs, implantable drug pump, etc) or pacemaker or implantable cardiac defibrillator
* Patient is a woman who is not using adequate contraception, is pregnant or breastfeeding or intends to become pregnant during the course of the study (a urine pregnancy test must be performed within 28 days prior to the Trial Lead Insertion Visit in women of child-bearing potential and the test result document)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kay Adair, Study Director — Boston Scientific Corporation
Locations (1):
- Hunter Pain Clinic, Newcastle, New South Wales, Australia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject was enrolled in this study.
Groups:
- Randomized: Eligible patients who were randomized in a 1:1:1:1:1:1 ratio to one of the six sequences of three treatment groups (sham stimulation, subthreshold spinal cord stimulation therapy 1, and subthreshold spinal cord stimulation therapy 2).
Period: First Intervention, 4 - 5 Days
Arm/Group | Randomized
Started | 1
Completed | 1
Not Completed | 0
Period: Second Intervention, 4 - 5 Days
Arm/Group | Randomized
Started | 1
Completed | 1
Not Completed | 0
Period: Third Intervention, 4 - 5 Days
Arm/Group | Randomized
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Randomized
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  Australia | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief
Description: Mean within-patient difference in average back pain intensity among treatment groups
Time Frame: 4,8,and 12 days post temporary lead(s) implantation
Population: No study data are available.
Arm/Group | Randomized
Number analyzed (Participants) | 0

2. Secondary Outcome: Pain Relief Responder Rate
Description: Difference in the proportion of subjects with ≥50% reduction in average back pain intensity among treatment groups
Time Frame: 4,8,and 12 days post temporary lead(s) implantation
Population: No study data are available.
Arm/Group | Randomized
Number analyzed (Participants) | 0

3. Secondary Outcome: Leg Pain Reduction
Description: Mean within-patient difference in average leg pain intensity among treatment groups
Time Frame: 4,8,and 12 days post temporary lead(s) implantation
Population: No study data are available.
Arm/Group | Randomized
Number analyzed (Participants) | 0

4. Secondary Outcome: Disability
Description: Mean within-patient difference in disability among treatment groups
Time Frame: 4,8,and 12 days post temporary lead(s) implantation
Population: No study data are available.
Arm/Group | Randomized
Number analyzed (Participants) | 0

5. Secondary Outcome: Percent Pain Relief
Description: Mean within-patient difference in overall percent pain relief among treatment groups
Time Frame: 4,8,and 12 days post temporary lead(s) implantation
Population: No study data are available.
Arm/Group | Randomized
Number analyzed (Participants) | 0

6. Secondary Outcome: Quality of Life, as Measured by EQ-5D-5L
Description: Mean within-patient difference in quality of life among treatment groups
Time Frame: 4,8,and 12 days post temporary lead(s) implantation
Population: No study data are available.
Arm/Group | Randomized
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: No study data are available
Arm/Group | Randomized
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes